CLINICAL TRIAL: NCT02106286
Title: The Influence of Beta-blockade on Cardiopulmonary Function Measured by Cardiopulmonary Exercise Testing
Brief Title: Effects of Beta-blockade on Cardiopulmonary Exercise Testing
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Michelle Mossa (Other Government)
Responsible Party: Sponsor-Investigator, Michelle Mossa, Research and Development Deputy Director, Liverpool University Hospitals NHS Foundation Trust
Organization: Liverpool University Hospitals NHS Foundation Trust (Other Government)
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 11/NW/0810
Record Dates: First submitted 2014-03-31; First posted 2014-04-08 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2014-04

CONDITIONS: Abdominal Aortic Aneurysm Patients Under Surveillance
Keywords: Cardiopulmonary exercise test; surgery; abdominal aortic aneurysm; anaerobic threshold; fitness; beta-blockers
MeSH Terms: conditions — Aortic Aneurysm, Abdominal | interventions — Bisoprolol

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bisoprolol (Active Comparator): Patients not betablocked at baseline receive an acute 72hr dose of beta blocker therapy before CPET
  Interventions: Drug: Bisoprolol
- No Bisoprolol (No Intervention): No beta blocker given

INTERVENTIONS:
Drug: Bisoprolol
  Arms: Bisoprolol

SUMMARY:
A major determinant of perioperative mortality is the inability of the heart to increase its output in response to surgical stress. This is termed perioperative cardiac failure (PCF), and may only be apparent postoperatively when oxygen demand is increased. The risk of perioperative cardiac complications is the summation of the individual patient's risk and cardiac stress related to the surgical procedure1. The functional capacity of the patient determines their ability to support the postoperative demand of increased oxygen consumption, and therefore of cardiac output. Exercise capacity is one of the most powerful predictors of cardiovascular and all cause mortality2. Cardiopulmonary exercise test (CPET) is an established investigation used, among other applications, in the preoperative assessment of patient fitness for surgery3. CPET involves monitoring the electrocardiographic trace and the exhaled gas mixture (particularly CO2, whose production depends on aerobic metabolism), during incremental exercise (usually on an exercise bike), on room air. Several parameters can be measured during CPET, including maximal systemic oxygen delivery, the anaerobic threshold (the oxygen delivery value at which anaerobic metabolism begins), maximum workload, and ST segment depression/elevation (as in a standard exercise tolerance test). The cardiopulmonary "performance" during CPET has been correlated with postoperative outcome3. Pulmonary function tests will be performed in order to assess lung function.

It is well known that therapy with beta-blockers in patients with ischaemic heart disease and cardiac failure reduces perioperative morbidity and mortality4-7. However, beta blockers reduce myocardial contractility and the heart rate response to adrenergic stimulation, thus blunting the physiological response to stress/surgery/exercise. Whilst this mechanism may protect the heart perioperatively, it may decrease the ability of some patients to withstand other complications. This potential decrease in "performance" has never been quantified.

There is no agreement on whether preoperative CPET should be performed on or off beta-blockers and, at Aintree in particular, it is standard procedure to take patients off beta-blockers prior to their CPET. Some argue that, as beta-blockade should be maintained in the perioperative period, CPET should be performed on medications, even if these could mask the presence significant ischaemic heart disease (a significant, modifiable, risk factor for surgery by beta blockade), and even if it is not always possible to maintain beta-blockade throughout the whole postoperative period. For these reasons, other clinicians prefer to perform CPET off beta-blockers, thus, potentially, overestimating the perioperative cardiorespiratory "performance", which may be diminished once the medications are resumed. Patients on long-term beta blockade may develop some tolerance to the medications, so the effect of acute and chronic beta blockade on cardiorespiratory performance may also be different.

Aim To compare cardiopulmonary performances on and off beta blockers as objectively assessed by cardiopulmonary exercise testing.

DETAILED DESCRIPTION:
Study design

We propose an interventional study investigating the effects of acute and chronic beta-blockade on cardiorespiratory performance prior to elective surgery.

We aim to recruit 64 abdominal aortic aneurysm (AAA) patients under surveillance who will undergo 2 cardiopulmonary exercise tests to investigate the effect of beta blockade on cardiopulmonary performance. This sample size is calculated by using a 2-tailed sample t-test, with 90% power to detect an estimated increase of 10% in oxygen delivery (VO2) at anaerobic threshold. We also estimated a drop-out rate of about 25% which is built into our power calculation estimates.

Interventions

Patients on long term beta blockade will be studied to investigate the effect of chronic beta blocker use. They will undergo two CPETs, the first on beta blockers, the second after discontinuing their beta blocker for at least 48 hours.

Patients not on beta blockers will be studied to investigate the effect of acute beta blockade. They will undergo two CPETs, the first off medication, the second after commencement of beta blockade (weight adjusted, started 48 hours prior to CPET).

Potential subjects will be provided with the patient information sheet in clinic, 1-2 weeks prior to their initial CPET. They will be given at least 1 week to consider the study in which the investigators will follow them up via a telephone call. Informed consent to participate in the study will be obtained at their initial (standard care) CPET.

All consenting subjects will perform exercise using electro-magnetically braked equipment during a ramped-incremental protocol in two different occasions. Prior to the tests full lung function tests will be performed by body plethysmography. The exercise tests will be performed with subjects wearing nose clips and breathing through a mouthpiece throughout the test. The initial cycling workload will be zero but will progressively increase at a rate of 10-15 Watts/min. After a resting period of 30 seconds and 2 minutes warm up subjects will stop when they can cycle no further. All gas exchange parameters will be measured and a metabolic cart, heart rate and oxygen saturation will be monitored at pre and post testing.

Subjects will also be asked to score their perceived breathlessness and leg fatigue using modified Borg scores every minute during exercise, and inspiratory capacity will be measured every minute during the exercise test.

At the end of this test, they will be given a date for the 2nd CPET and a prescription for oral bisoprolol once daily (dose adjusted to patients body weight), to be started 48 hours prior to the test (two doses in total). Patients will be informed of potential side effects of the medications at this visit. This will be weight adjusted with a specific dose as follows: 1.25 mg if patent weighs 50-75 kg, 2.5 mg if 75-100 kg and 3.75 mg if >100 kg.

Patients will then attend for the 2nd CPET, following which bisoprolol will be discontinued or continued based on clinical indication.

If patients are already chronically on a beta blocker, they will have their first CPET while on medication, and then will be asked to stop the medication for a period of 48 hours before the second CPET. It is standard procedure to take the patient off beta blockers prior to their CPET at Aintree University Hospital. Patients will be informed of potential risks of stopping their beta blocker at their first visit. The beta blocker will be restarted or discontinued based on clinical indication after the second CPET.

ELIGIBILITY:
Inclusion Criteria:

1. >18 years of age inclusive, undergoing major surgery who are already on therapy with beta blockers
2. >18 years of age, undergoing major surgery who are not on beta blockers
3. Patient able to consent to study protocol
4. Ability to perform CPET on an exercise bike
5. AAA patients under surveillance.

Exclusion Criteria:

1. Known contraindication to bisoprolol (known intolerance, asthma or history of bronchospasm, II or III degree heart block, treatment with verapamil or ivrabadine, sinus bradycardia, Prinzmetal's angina),
2. Severe ischaemic heart disease (including acute coronary syndrome within 3 months of recruitment),
3. Inability to use an exercise bike
4. Stage IV and V chronic kidney disease
5. Uncontrolled hypertension
6. Patients withholding informed consent
7. Patients unable to give informed consent due to mental incapacity
8. Patients who find uncomfortable and anxiety provoking performing an exercise test
9. Patients who present contraindications (relative/absolute) to their first initial CPET based on the American Thoracic Society (ATS) exercise testing guidelines.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2011-02; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change in oxygen uptake | Baseline and 72hours post beta-blockade

CONTACTS AND LOCATIONS:
Locations (1):
- Aintree University Hospitals, Liverpool, United Kingdom

REFERENCES:
- [Derived] Key A, Parry M, West MA, Asher R, Jack S, Duffy N, Torella F, Walker PP. Effect of beta-blockade on lung function, exercise performance and dynamic hyperinflation in people with arterial vascular disease with and without COPD. BMJ Open Respir Res. 2017 Apr 5;4(1):e000164. doi: 10.1136/bmjresp-2016-000164. eCollection 2017. PMID 28409004
- [Derived] West MA, Parry M, Asher R, Key A, Walker P, Loughney L, Pintus S, Duffy N, Jack S, Torella F. The Effect of beta-blockade on objectively measured physical fitness in patients with abdominal aortic aneurysms--A blinded interventional study. Br J Anaesth. 2015 Jun;114(6):878-85. doi: 10.1093/bja/aev026. Epub 2015 Feb 24. PMID 25716221